CLINICAL TRIAL: NCT06117657
Title: Safety and Efficacy Clinical Study of KL-HIV-Tri01 in the Treatment of HIV Infected Subjects
Status: Unknown | Phase: Early Phase 1 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Affiliated Hospital of Guangdong Medical University (Other)
Responsible Party: Principal Investigator, Honghua He, Associated chief physician, Affiliated Hospital of Guangdong Medical University
Allocation: Not Applicable | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: CP-Tri01-001/01
Record Dates: First submitted 2023-10-31; First posted 2023-11-07 (Actual); Last update posted 2023-11-08 (Actual); Status verified 2023-11

CONDITIONS: HIV Infections
MeSH Terms: conditions — HIV Infections

STUDY DESIGN:
Intervention Model Description: Low dose group will be administrated with 2.4×10^11 vg/kg; Middle dose group will be administrated with 8.0×10^11 vg/kg; High dose group will be administrated with 2.4×10^12 vg/kg;
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- KL-HIV-Tri01 injection solution (Experimental): Subjects will be dosed with three different dose of KL-HIV-Tri01 injection solution at 2.4x10^11 vg/kg to 2.4x10^12 vg/kg.
  Interventions: Drug: Low dose KL-HIV-Tri01; Drug: Middle dose KL-HIV-Tri01; Drug: High dose KL-HIV-Tri01

INTERVENTIONS:
Drug: Low dose KL-HIV-Tri01 — Subjects will be dosed with single dose of KL-HIV-Tri01 at 2.4x10^11 vg/kg.
  Other Names: rAAV vector
Drug: Middle dose KL-HIV-Tri01 — Subjects will be dosed with single dose of KL-HIV-Tri01 at 8.0x10^11 vg/kg.
  Other Names: rAAV vector
Drug: High dose KL-HIV-Tri01 — Subjects will be dosed with single dose of KL-HIV-Tri01 at 2.4x10^12 vg/kg.
  Other Names: rAAV vector

SUMMARY:
This is an open- label, non- randomized, uncontrolled, dose-escalation pilot study to evaluate the safety and efficacy of KL-HIV-Tri01 injection solution in HIV infected subjects treated with HAART.

DETAILED DESCRIPTION:
This is an open- label, non- randomized, uncontrolled, dose-escalation pilot study to evaluate the safety and efficacy of KL-HIV-Tri01 injection solution expressing triple targets antibodies with broad HIV-1 neutralizing activity in HIV-1 infected adults on anti-retroviral therapy (ARV). Nine subjects will be enrolled and administered with three different doses of KL-HIV-Tri01. Subjects will provide informed consent and then undergo screening assessments up to 1 month prior administration of KL-HIV-Tri01. All subjects will undergo 52 weeks safety observation and will be encouraged to enroll in an extension study to evaluate long- term safety of KL-HIV-Tri01 for total 5 years.

ELIGIBILITY:
Inclusion Criteria:

1.18 (not inclusive) to 80 (inclusive) years of age, both male and female.

2. Conform to the Chinese AIDS Diagnosis and Treatment Guidelines (2021), HIV positive, and received HAART treatment for ≥ 3 months before enrollment.

3. CD4+T cell count≥500 cells/μl.

4. On a stable antiretroviral regimen before enrollment and viral load less than 40 copies/mL in two consecutive tests one year prior to enrollment.

5. Willing to fully understand the purpose, nature, method, and potential adverse reactions that may occur during the discontinuation period of the experiment, voluntarily participate in this experiment and sign an informed consent form.

Exclusion Criteria:

1. Bleeding disorder diagnosed by a doctor (e.g. factor deficiency, coagulopathy, or platelet disorder requiring special precautions) or significant bruising or bleeding difficulties with IM injections or blood draws.
2. Active viral infections, such as HBV, HCV, CMV, or other viruses that the investigator believes will affect clinical research.
3. Any opportunistic infection in the past one year, such as tuberculosis, cryptococcosis, which is not cured after treatment.
4. Currently treated with Immunosuppressive medications or steroids.
5. Previous receipt of HIV vaccine, antibody or gene therapy.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 9 (Estimated)
Dates: Start 2023-11-10 (Estimated); Primary Completion 2024-08-20 (Estimated); Study Completion 2025-09-10 (Estimated)

PRIMARY OUTCOMES:
Number and severity of AEs and SAEs | Day 0 through 52 Weeks after KL-HIV-Tri01 administration
  AEs and SAEs from the date of product administration will be recorded through the last study visit. The relationship between AEs and the study product was assessed by the investigator based on clinical judgment and the definitions outlined in the protocol.
Neutralizing Antibodies Against KL-HIV-Tri01 Capsid | Day 0 through 52 Weeks after KL-HIV-Tri01 administration
  Anti-KL-HIV-Tri01 Capsid antibodies were analyzed by enzyme-linked immunosorbent assay (ELISA) using a vector-matched AAV capsid as the capture agent.
Inhibitors of broadly neutralizing antibodies | Day 0 through 52 Weeks after KL-HIV-Tri01 administration
  Inhibitors against broadly neutralizing antibodies expressed by KL-HIV-Tri01 were analyzed by enzyme-linked immunosorbent assay (ELISA) .
Cells mediated immune response against capsids and bNabs | Day 0 through 52 Weeks after KL-HIV-Tri01 administration
  Number of participants with T-cell response to AAV capsid and transgene products was planned to be reported.

SECONDARY OUTCOMES:
Concentration and titer of serum neutralizing antibodies | Day 0 through 52 Weeks after KL-HIV-Tri01 administration
  The serum concentration and titer of neutralizing antibodies produced by KL-HIV-Tri01 at specified time intervals for 52 weeks after dosing was determined
CD4+T, CD8+T cell count | Day 0 through 52 Weeks after KL-HIV-Tri01 administration
  The clinical effects of KL-HIV-Tri01 on CD4+T and CD8+T cell count were assessed. CD4+T and CD8+T Cell Count (cells/mL) shown as reported by the Clinical Center serology lab
viral load | Day 0 through 52 Weeks after KL-HIV-Tri01 administration
  The clinical effects of KL-HIV-Tri01 on viral load were assessed after interruption of HAART.
Time to interrupt HAART treatment | Day 0 through 52 Weeks after KL-HIV-Tri01 administration
  The duration of anti-HIV replication effection of the neutralizing antibodies produced by KL-HIV-Tri01were assessed after interruption of HAART.

CONTACTS AND LOCATIONS:
Overall Officials: Honghua He, MD, Principal Investigator — Affiliated Hospital of Guangdong Medical University

IPD SHARING:
Plan to Share IPD: No